CLINICAL TRIAL: NCT06954090
Title: SIGNAL - Body Fluid Proteome SIGnatures for persoNALised Intervention to Prevent Cardiovascular and Renal Complications in Diabetes
Brief Title: Urinary Proteomics to Guide Early Intervention to Prevent Complications in Type 2 Diabetes - a Feasibility Study
Acronym: SIGNAL
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Mosaiques Diagnostics GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-518682-95; 2024-518682-95-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-14; First posted 2025-05-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Type 2 DM; Type 2 DM /Diabetic Nephropathy; Albuminuria
Keywords: urine proteomics; precision medicine; prevention of diabetic complications; personalized treatment; biomarker; CKD273
MeSH Terms: conditions — Albuminuria | interventions — semaglutide; finerenone; dapagliflozin

STUDY DESIGN:
Intervention Model Description: Low intervention feasibility study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Semaglutide (Active Comparator): 3 urine proteomic risk scores will be measured in the study. The CKD273 urine proteomic risk score, a well-established tool used to predict the risk of chronic kidney disease (CKD) progression, CAD160 urine proteomic risk score to predict the risk of coronary artery disease (CAD) and HF2 urine proteomic classifier to predict the risk of heart failure (HF).
  In addition a Support Vector Machine (SVM), a supervised machine learning algorithm will perform in silico treatment simulations and calculate the change in classification scores for 3 different potential interventions: GLP1-RA semaglutide, SGT2-i dapagliflozin and GLP1-RA finerenone. Based on these changes (with the largest beneficial change indicating the most effective treatment), the most suitable intervention can be selected and the participent will be allocated.
  Interventions: Drug: Semaglutide, 1.34 mg/mL
- Finerenone (Active Comparator): 3 urine proteomic risk scores will be measured in the study. The CKD273 urine proteomic risk score, a well-established tool used to predict the risk of chronic kidney disease (CKD) progression, CAD160 urine proteomic risk score to predict the risk of coronary artery disease (CAD) and HF2 urine proteomic classifier to predict the risk of heart failure (HF). In addition a Support Vector Machine (SVM), a supervised machine learning algorithm will perform in silico treatment simulations and calculate the change in classification scores for 3 different potential interventions: GLP1-RA semaglutide, SGT2-i dapagliflozin and GLP1-RA finerenone. Based on these changes (with the largest beneficial change indicating the most effective treatment), the most suitable intervention can be selected and the participent will be allocated.
  Interventions: Drug: Finerenone Oral Tablet
- Dapagliflozin (Active Comparator): 3 urine proteomic risk scores will be measured in the study. The CKD273 urine proteomic risk score, a well-established tool used to predict the risk of chronic kidney disease (CKD) progression, CAD160 urine proteomic risk score to predict the risk of coronary artery disease (CAD) and HF2 urine proteomic classifier to predict the risk of heart failure (HF). In addition a Support Vector Machine (SVM), a supervised machine learning algorithm will perform in silico treatment simulations and calculate the change in classification scores for 3 different potential interventions: GLP1-RA semaglutide, SGT2-i dapagliflozin and GLP1-RA finerenone. Based on these changes (with the largest beneficial change indicating the most effective treatment), the most suitable intervention can be selected and the participent will be allocated.
  Interventions: Drug: Dapagliflozin (DAPA)

INTERVENTIONS:
Drug: Semaglutide, 1.34 mg/mL — Semaglutide will be introduced at a dose of 0.25 mg/week subcutaneous injection, escalated to 0.5 and 1.0 mg/week after 4 and 8 weeks if tolerated.
  Other Names: Ozempic
  Arms: Semaglutide
Drug: Finerenone Oral Tablet — Finerenone will be introduced at a dose of 10 mg/day in patients with a serum potassium level < 4.8 mmol/l and eGFR < 60 ml/min/1.73 m2 and escalated to 20 mg/day after 4 weeks if the serum potassium level is still < 4.8 mmol/l. Starting dose is 20 mg/day if eGFR ≥ 60 ml/min/1.73 m2. The dosage will be reduced or discontinued in patients who develop hyperkalemia (serum potassium > 5.5 mmol/l).
  Arms: Finerenone
Drug: Dapagliflozin (DAPA) — Dapagliflozin will be introduced at a dose of 10 mg/day. The dose can be reduced at any time during the trial if required by the subject's tolerance to the product.
  Arms: Dapagliflozin

SUMMARY:
Title:

Body fluid proteome SIGnatures for persoNALised intervention to prevent cardiovascular and renal complications in diabetes.

Aim:

To explore the feasibility of using urinary proteomic risk scores in clinical practice to identify patients at risk of developing end organ damage and identify which patients should receive additional renocardiovascular protective treatment.

DETAILED DESCRIPTION:
Background:

Diabetes and its associated complications impose a significant burden on both patients and societies. Despite advancements in lowering blood glucose, the elevated risk of developing cardiovascular disease (CVD) and chronic kidney disease (CKD) remains a pressing concern, underscoring the need for optimized prevention strategies and improved therapeutic options. Recent developments in glucose-lowering drugs, such as sodium-glucosecotransporter- 2-inhibitors (SGLT2-i) and glucagon-like-peptide-1 receptor agonists (GLP1-RA), as well as the use of the non-steroidal mineralocorticoid receptor antagonist (nsMRA) finerenone, have shown promising cardiovascular and renal protection. Currently, there is no reliable method for predicting personalized treatment responses in diabetic complications. Consequently, benefits of treatment are under dispute, due to a large number of patients not responding. The use of SGLT2-i, nsMRA and GLP1-RA in CKD has happened largely in parallel, all agents have demonstrated benefit, but it is not yet clear how to prioritize between the drugs or if all should be combined. This study builds upon previous scientific work that have investigated the urine proteome and identified several biomarkers able to predict early diabetes associated complications.

CKD273 urine proteomic risk score is a well-established tool used to predict the risk of chronic kidney disease (CKD) progression. CAD160 is urine proteomic risk score to predict the risk of coronary artery disease (CAD). HF2 urine proteomic classifier is used to predict the risk of heart failure (HF).

Urine sample analysis is based on capillary electrophoresis coupled with mass spectrometry (CE-MS) to determine these risk scores.

Urine proteomic scores are continous numerical values. Higher score means that the urinary peptide pattern is more similar to that of patients with progressive disease. A lower score indicates a peptide profile more typical of healthy individuals.

In addition a Support Vector Machine (SVM), a supervised machine learning algorithm will perform in silico treatment simulations and calculate the change in classification scores for 3 different potential interventions: GLP1-RA semaglutide, SGT2-i dapagliflozin and GLP1-RA finerenone. Based on these changes (with the largest beneficial change indicating the most effective treatment), the most suitable intervention can be selected and the participent will be allocated.

Design:

Single-centre, open-label, parallel group (intervention group) with 6 months intervention.

Population:

Type 2 diabetes without history of heart failure NYHA Class IV or advanced diabetic kidney disease with an estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1.73m2 or urinary albumin creatinine ratio (UACR) > 200 mg/g.

Objectives:

To assess the feasibility of using proteomic classifiers in clinical practice for response prediction in a prospective study. We will use urinary proteomic classifiers: CKD273, CAD160 and HF2 to identify patients suited for additional medical treatment with sodium-glucose-cotransporter-2 (SGLT2)- inhibitors, glucagon-like-peptide-1 GLP-1 receptor agonists or non-steroidal mineralocorticoid receptor antagonist.

Interventions:

The SGLT2 inhibitor dapagliflozin 10 mg daily, the nsMRA finerenone 10-20 mg daily, and the GLP-1 receptor agonist semaglutide 0.25-1.0 mg once weekly. The medication will be given stepwise according to a prespecified algorithm and guided by the response on UACR.

Endpoints:

Primary endpoint is feasibility of using urinary proteomic classifiers in clinical practice, while secondary endpoints are changes in UACR and urinary proteomic signatures after 6 months of treatment.

Time schedule:

The study is expected to start inclusion June 1st 2025. The recruitment period is 6 months, the intervention period is 6 months and hence the study is expected to be terminated May 31st 2026.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age.
2. Type 2 diabetes with no clinical signs of HF NYHA Class IV
3. Able to understand the written participant information and give informed consent.

Exclusion Criteria:

1. Heart failure NYHA class IV at screening
2. Moderately - or severely increased albuminuria with a UACR ≥ 200 mg/g or CKD with an eGFR < 30 ml/min/1.73m2 at the screening visit.
3. A female who is pregnant, breastfeeding, or intends to become pregnant, or women of childbearing potential (WOCBP) who are not using highly effective contraceptive methods.
4. Receiving therapy with all three of the study medication prior to enrolment.
5. Myocardial infarction, unstable angina, stroke, or transient ischemic attack within 12 weeks prior to enrolment
6. Known or suspected hypersensitivity to the study medications or related products
7. History of pancreatitis at the screening visit
8. Body mass index < 18.5 kg/m2 at the screening visit
9. Type 1 diabetes
10. Serum potassium > 5.0 mmol/L at the screening visit
11. Addison's Disease
12. Concomitant treatment with strong CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, ritonavir, nelfinavir, cobicistat, clarithromycin, telithromycin, nefazodone)
13. Treatment with a potassium-sparing diuretic (amiloride, triamterene)
14. Treatment with other mineralocorticoid receptor antagonist than finerenone (e.g., spironolactone, eplerenone, esaxerenone, canrenone)
15. Elevated Alanine Aminotransferase (ALT) > 3x upper normal limit, autoimmune hepatitis, and/or severe hepatic impairment (including but not limited to a history of hepatic encephalopathy, a history of oesophageal varices or a history of portocaval shunt.)
16. Autosomal dominant or autosomal recessive polycystic kidney disease
17. Lupus nephritis or ANCA-associated vasculitis, or any other primary or secondary kidney disease requiring immunosuppressive therapy within 6 months prior to screening
18. Kidney transplant or dialysis
19. Presence or history of malignant neoplasms (except basal cell skin cancer or squamous cell skin cancer) within five years before screening.
20. Any other history, condition, therapy, or uncontrolled intercurrent illness that could, as judged by the investigator, affect participant safety or compliance with study requirements.
21. Known or suspected abuse of narcotics.
22. Participant in another intervention study,
23. Vulnerable (i.e., under guardianship) or mentally incapacitated subjects (i.e., not able to understand and sign the informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility for this study is based on gender identity, not biological sex. This means that the study is open to anyone who identifies as male or female, regardless of their biological sex. We recognize and respect each person's gender identity, and eligibility is determined by how they identify.
Enrollment: 50 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Proteomic feasibility | 2 weeks from sampling
  Achieve urine proteomic results within 2 weeks of sampling for at least 90% of the participants in clinical practice.
Evaluation of medical treatment | 3 weeks from sampling
  Ensure that urine proteomic results are interpreted for evaluating medical treatment in at least 90% of participants.

SECONDARY OUTCOMES:
Urine Albumin-to-Creatinine Ratio | Over the 6 month of the follow up from screening visit to the end of study.
  Changes in UACR from screening visit to the end of study
Urinary proteomic signatures | Over the 6 month of the follow up from screening visit to the end of study.
  Changes in urinary proteomic signatures from screening visit to the end of study:
  Urine proteomic risk scores are continous numerical values. Higher score means urinary peptide pattern is more similar to that of patients with progressive disease. A lower score indicates a peptide profile more typical of healthy individuals.
  CKD273, CAD160 and HF2 urine proteomic risk-scores and their changes will be measured from urine samples during the study.

OTHER OUTCOMES:
Assessment of health economics | 6 months from all participent data is collected
  Potential adoption of biomarkers in clinical practice for patient stratification requires the evaluation of cost-effectiveness compared to current gold standards.
  During he cost effectiveness analysis, health economic modelling will be performed to translate implementation of the molecular predictors into quantitative estimates of clinical and economic benefits and costs incomparison to the standard of care. Markov models will be developed using specialized software (TreeAge Healthcare Pro software, Williamstown, USA) and incremental cost-effectiveness ratios (ICER) will be calculated. The analysis will be conducted and reported according to CHEERS Statement.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, Clinical Professor, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Hajdú-Bihar, Denmark

IPD SHARING:
Plan to Share IPD: No